CLINICAL TRIAL: NCT03112551
Title: Safety and Efficacy of Twelve Hours Duration of Magnesium Sulphate in the Treatment of Eclampsia in Low Resource Setting in Sudan
Brief Title: Safety and Efficacy of Twelve Hours Duration of MgSO4 in the Treatment of Eclampsia in Low Resource Setting in Sudan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Gadarif University (Other)
Responsible Party: Principal Investigator, AbdelAziem AbdAllah Ali, Prof., Gadarif University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GadarifU
Record Dates: First submitted 2017-03-28; First posted 2017-04-13 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2017-11

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group 1 (Active Comparator): group one will be treated with 24 hours maintenance dose of magnesium sulphate
  Interventions: Drug: Adminstration of magnesium Sulphate for treatment of eclampsia
- group 2 (Experimental): group 2 will be treated with 12 hours maintenance dose of magnesium sulphate
  Interventions: Drug: Adminstration of magnesium Sulphate for treatment of eclampsia

INTERVENTIONS:
Drug: Adminstration of magnesium Sulphate for treatment of eclampsia — A total of 100 eclamptic patients are suspected to be approached alternately and subcategorized into two groups - one group will be treated with 24 hours maintenance dose of magnesium sulphate (Group-1; n=50), and the other with 12 hours maintenance dose of magnesium sulphate (Group-2; n=50).

SUMMARY:
the investigators assume that magnesium sulphate for treating eclampsia can be safely reduced from 24 hours to shorter duration of therapeutic anticonvulsant effect for 12 hours. Short duration of drug exposure is suitable for low resource setting where there is little tools or busy staff for monitoring drug toxicity.

DETAILED DESCRIPTION:
The idea of using 12 hours duration of magnesium sulphate for treating eclampsia may be effective and attractive, especially in settings with limited resources and where there is no availability of tools to monitor the serum level of magnesium sulphate. This is because the most common reported maternal adverse effects of magnesium sulphate are minor and may be confused with other symptom of eclampsia of even labor.The administration of Magnesium sulphate for 24 hours in the absence of monitoring of the serum magnesium sulphate might be life threatening in a resource- challenged situation , thus the current study is planned to be conducted to investigate the efficacy and safety of shorter duration (12 hours) of magnesium sulphate therapy in preventing development of convulsions in cases of eclampsia.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of eclampsia
* must accept to participate in the study

Exclusion Criteria:

* epilepsy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients who will receive magnesium sulfate and develop drug toxicity | 12 - 24 hours
  the adverse effect of magnesium sulphate either minor signs:flushing, increased warmth and sweating, nausea, vomiting, headaches, muscle weakness and blurred vision or major effects such as absent tendon reflexes and oliguria.

CONTACTS AND LOCATIONS:
Locations (1):
- Gadarif University, Gedaref, Sudan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diaz V, Long Q, Oladapo OT. Alternative magnesium sulphate regimens for women with pre-eclampsia and eclampsia. Cochrane Database Syst Rev. 2023 Oct 10;10(10):CD007388. doi: 10.1002/14651858.CD007388.pub3. PMID 37815037